CLINICAL TRIAL: NCT04677478
Title: Impact of the Respiratory Isolation on the Quality of Life in Patients Hospitalized for Tuberculosis or COVID-19
Acronym: ISO-BK
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200227
Record Dates: First submitted 2020-12-15; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-12

CONDITIONS: Tuberculosis; Covid19
MeSH Terms: conditions — Tuberculosis; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Impact of respiratory isolation on quality of life — Semi-structured interviews

SUMMARY:
The respiratory isolation could have a harmful impact on the well-being of patients, especially in a psychological point of view such as anxiety and depression disorders or through the relationship with medical team and/or relatives but also in terms of informations.

The evaluation of the impact of respiratory isolation in patients hospitalized for tuberculosis or COVID-19 could allow to identify the different kinds of problems encountered by these patients (physical, psychological, sociological, informations, ...) in order to adapt the environment for efficient care and to improve patient's well-being.

The purpose of this research is to evaluate the psychological impact of the respiratory isolation on the quality of life in patients hospitalized for tuberculosis or COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who are more than 18 years old hospitalized in respiratory isolation for tuberculosis or COVID-19.
2. Patient able to understand questions and to communicate verbally with investigators.
3. Patient who has given his consent.

Exclusion Criteria:

1. Patient deprived of their rights
2. Patient under tutorship or guardianship or under the protection of a conservator
3. Tuberculosis without respiratory isolation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for tuberculosis or COVID-19 and placed in respiratory isolation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
Quality of life using semi-structured interview. | at 28 days respiratory isolation
  Quality of life will be assessed using semi-structured interview.
Quality of life using 36-Item Short Form Health Survey (SF-36) | at 28 days respiratory isolation
  Quality of life will be assessed using SF-36. SF-36 is a set of generic, coherent, and easily administered quality-of-life measures. These measures rely upon patient self-reporting. Items are grouped into three categories: functional status, well-being, overall health assessment. The scores for the different items are coded and then summed and transformed linearly on a scale ranging from 0 to 100.
Quality of life using State-Trait Anxiety Inventory (STAY) A+B scale | at 28 days respiratory isolation
  The State-Trait Anxiety Inventory is a self-rated scale. Each type of anxiety has its own scale of 20 different questions that are scored. STAY-YA and STAY-YB Scores range from 20 to 80. A higher score is higher anxiety.
Quality of life using Beck Depressive Inventory (BDI) -13 | at 28 days respiratory isolation
  It is a self-rated scale. each item is made up of 4 sentences corresponding to 4 degrees of intensity of increase in a symptom: from 0 to 3. The overall score is obtained by adding the scores of the 13 items. The range of the scale is 0 to 39.

IPD SHARING:
Plan to Share IPD: Undecided